CLINICAL TRIAL: NCT00246558
Title: Is There a Connection Between a Tight Achilles Tendon, Hyperpronation of the Foot and Pain in the Anterior Part of the Knee
Brief Title: Tight Achilles Tendon, Hyperpronation and Anterior Knee Pains
Status: Withdrawn | Type: Observational
Why Stopped: The study stopped due to unforeseen circumstances.
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-02-011-OSi
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Tight Achilles Tendon; Hyperpronation of the foot
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to investigate the prevalence of pain in the anterior part of the knee, amongst youngsters between 16 and 18 years of age.

Furthermore, this trial intends to study the connection between the pain, hyperpronation of the foot and tight Achilles tendon.

We want to find out if there is a need of an early effort in terms of information, training and/or support for the shoes.

DETAILED DESCRIPTION:
All students (around 300) between 16 and 18 years of age from one Gymnasium, receives a questionnaire. They are asked to answer whether they have had pain in the anterior part of their knee within the last month. If so they are invited to participate in a scientific study. An equivalent group with no pain are invited to participate as a control group.

In both groups navicular drop and drift will be measured together with the dorsal flexion. The investigations are made single-blinded as the investigators do not know if the "patient" has pain or not.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, and for those being under 18 years of age, their parents signature.
* Anterior knee pain syndrome and for the control group: no knee pain syndrome

Exclusion Criteria:

* Former knee surgery
* Any form of arthritis
* Diagnosed meniscus or other injuries in the knee

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Ole Simonsen, MD, Principal Investigator — Northern Orthopaedic Division, Denmark
Locations (1):
- Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland, Denmark